CLINICAL TRIAL: NCT03025529
Title: Transcranial Stimulation for Essential Tremor
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Investigator leaving institution
Sponsor: Beth Israel Deaconess Medical Center (Other)
Responsible Party: Principal Investigator, Ludy Shih, Assistant Professor of Neurology, Beth Israel Deaconess Medical Center
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Device Feasibility
Other Study IDs: 2015P000011
Record Dates: First submitted 2017-01-06; First posted 2017-01-19 (Estimated); Last update posted 2017-12-19 (Actual); Status verified 2017-12

CONDITIONS: Essential Tremor
MeSH Terms: conditions — Essential Tremor | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Intervention Model Description: This is a crossover design with two groups, preceded by a separate single group of healthy controls in a pilot study to assess feasibility of obtaining the cerebellocortical inhibition measure
Masking Description: In the single group pilot study, there is no intervention and no masking-- just obtaining an MRI and a cerebellocortical inhibition measure. There were 8 subjects in this phase of the study. There were no subjects enrolled in the crossover design phase of this study.
Oversight: Data Monitoring Committee: No

ARMS (3):
- Active Cerebellar rTMS (Experimental): Cerebellar rTMS will be carried out in ET subjects using a MagPro stimulator with a double cone coil at 1Hz (1 pulse every second) for 3 minutes on the left and 3 minutes on the right, at the cerebellar location indicated by resting state functional connectivity MRI analysis. Subjects with ET will undergo 5 consecutive daily sessions of cerebellar rTMS at either the connectivity map generated target or sham rTMS and then crossover to the other target after 2 weeks. Subjects will be blinded to the treatment order assignment. The intensity of the stimulation will be determined as 90% of the resting motor threshold, to be determined at the beginning of the first visit.
  Interventions: Device: Transcranial Magnetic Stimulation
- Sham Cerebellar rTMS (Sham Comparator): In sham rTMS, the same parameters and procedures as Treatment Procedures 4-8 will be used, except that the coil will be angled 90 degrees from the scalp, resting on one wing of the coil.
  Interventions: Device: Sham Transcranial Magnetic Stimulation
- Healthy control pilot (No Intervention): This pilot phase is done to assess feasibility of obtaining MRI and cerebellocortical inhibition measures in healthy control subjects.

INTERVENTIONS:
Device: Transcranial Magnetic Stimulation — Transcranial Magnetic Stimulation or TMS is a noninvasive procedure (meaning it does not enter the body) that is used to stimulate a part of the brain using a magnetic field. This magnetic field can pass through the head safely and painlessly. TMS can be used to change activity in the brain.
  Other Names: TMS
  Arms: Active Cerebellar rTMS
Device: Sham Transcranial Magnetic Stimulation — Sham Transcranial Magnetic Stimulation or sham TMS is like active TMS, a noninvasive procedure (meaning it does not enter the body) that is used to stimulate a part of the brain using a magnetic field. TMS can be used to change activity in the brain but in this intervention, the coil will be angled 90 degrees from the scalp, resting on one wing of the coil, and therefore will not be delivering active TMS.
  Other Names: Sham TMS
  Arms: Sham Cerebellar rTMS

SUMMARY:
The main purpose of this study is to see if transcranial magnetic stimulation (TMS) can be used to help study brain function in healthy people and in those with neurological diseases like essential tremor. This portion of the study is being done to establish the optimal methods for stimulating the brain to measure its responses.

DETAILED DESCRIPTION:
Essential tremor (ET) is a movement disorder characterized by tremor of both hands, and often head and voice, affecting approximately 4.8-6.7 million individuals over the age of 40 in the United States alone. Hand tremor can limit basic activities of daily living like feeding, drinking, writing and dressing. While medications can be effective for tremor, they are often poorly tolerated due to their sedative or neuronal activity depressant properties. Surgical options such as deep brain stimulation of the ventral intermedius thalamus (Vim DBS) can be highly effective but its invasive nature limits its popularity. Noninvasive brain stimulation has demonstrated the ability to reduce tremor but precisely where to target brain stimulation to achieve the best results is currently unknown.

Repetitive transcranial magnetic stimulation (rTMS) enables noninvasive, selective and sustained modulation of specific neural networks, and can lead to clinical benefits in debilitating neurologic and psychiatric disorders, including medication-resistant depression, paresis following stroke or traumatic brain injury, Parkinson's disease, or dementia. There is also recent evidence that rTMS of the cerebellum can relieve hand tremor due to essential tremor. TMS uses electromagnetic induction to generate controlled currents in targeted brain structures that can be identified and defined using MRI-based neuronavigation. TMS is safe if appropriate guidelines are adhered to. To date, the impact of rTMS on ET has not been sufficiently established, but pilot studies offer promising results.

The investigators are testing whether MRI-guided neuronavigated cerebellar paired pulse TMS demonstrates abnormal physiologic measures in ET subjects compared to controls and whether there is reduction of tremor via cerebellar rTMS in patients with ET. The investigators plan to collect imaging, functional and neurophysiological assessments before and after the rTMS to identify the mechanistic underpinnings of rTMS-induced changes in tremor and cerebello-cortical inhibition.

ELIGIBILITY:
Inclusion Criteria for ET subjects:

1. Outpatients with essential tremor as diagnosed and confirmed by movement disorder specialist
2. Women of child-bearing potential must provide a negative pregnancy test at entry into the study
3. Stable doses of all medications for at least 14 days prior to study entry and for the duration of the study,
4. At least a 1cm amplitude tremor as judged by the screener using a ruler

Inclusion Criteria for Healthy Volunteers:

1. Healthy subjects without tremor and without significant neurologic disease suggestive of cerebellar ataxia or other neurodegenerative diseases
2. Ages 18-80

Exclusion Criteria:

1. Any unstable illness or concomitant medical condition that, in the investigator's opinion, precludes participation in this study, including disorders that may affect gait or balance (i.e., stroke, arthritis, etc).
2. Pregnancy or lactation.
3. Concurrent participation in another clinical study.
4. Dementia or other psychiatric illness that prevents the patient from giving informed consent (Montreal Cognitive Assessment Score score less than or equal to 21).
5. Legal incapacity or limited legal capacity.
6. Tremor derived from any cause other than essential tremor (Parkinson's disease, drug-induced, anxiety-induced) in the clinical assessment at screening
7. Currently taking lithium or amiodarone or any other drug judged to be contributing to tremor as judged by the investigator (may be a cause of tremor)
8. No medication is an absolute exclusion from TMS. Medications will be reviewed by the responsible MD and a decision about inclusion will be made based on the following:

   * The patient's past medical history, drug dose, history of recent medication changes or duration of treatment, and combination with other Central Nervous System active drugs.
   * The published TMS guidelines review of medications to be considered with TMS
9. History of seizures, diagnosis of epilepsy, history of abnormal (epileptiform) EEG, or family history of treatment resistant epilepsy with the exception of a single seizure of benign etiology (e.g. febrile seizures) in the judgement of the investigator
10. TMS and MRI-Specific exclusion criteria including:

    * Known metal in the head (such as a surgical aneurysm clip) or a history of prior neurosurgical procedures.
    * Ferromagnetic bioimplants activated by any electronic, mechanical or magnetic means, such as cochlear implants, pacemakers, medication pumps, vagal stimulators, deep brain stimulators, neurostimulators, biostimulators, or ventriculo-peritoneal shunts.
    * Subjects who have or might have bullet fragments or other shrapnel (veterans or workers exposed to metal in their work environment).
    * Subjects with metallic paint (e.g. color contact lenses, tattoos, metallic eyeliner)
    * Subjects expressing significant claustrophobia.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2015-02; Primary Completion 2016-11-28 (Actual); Study Completion 2016-11-28 (Actual)

PRIMARY OUTCOMES:
Tremor Reduction | One week after intervention
  tremor rating scale with questions regarding impact of tremor on activities of daily living and an physician-rated assessment of degree of tremor in hands, head, voice, and while drawing and writing

SECONDARY OUTCOMES:
Cerebellocortical Inhibition | One week after intervention
  Ratio of conditioned to unconditioned motor evoked potentials

CONTACTS AND LOCATIONS:
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States